CLINICAL TRIAL: NCT06801145
Title: The Effect of Video-supported Education About the Intensive Care Process on Anxiety Levels and the ICU Experience of Patients Scheduled for Open-heart Surgery
Brief Title: The Effect of Video-supported Education on Anxiety Levels and the ICU Experience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeynep Turak (Other)
Responsible Party: Sponsor-Investigator, Zeynep Turak, Master student, Ataturk University
Organization: Ataturk University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: B.30.2.ATA.0.01.00/363
Record Dates: First submitted 2024-04-10; First posted 2025-01-30 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Open Heart Surgery
Keywords: BYPASS; OPEN HEART SUNGERY; Anxiety; patient education; intensive care experience
MeSH Terms: conditions — Anxiety Disorders | interventions — Educational Status; Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Video training will be provided 48 hours before the surgery.
  Interventions: Other: Education with Video
- Control group (No Intervention): This group will receive no intervention other than the applied scales; only standard nursing care will be maintained.

INTERVENTIONS:
Other: Education with Video — Patients in the experimental group will be trained by the researcher 48 hours before the surgery with a video providing information about the intensive care process.
  Arms: Experimental group

SUMMARY:
This study was conducted to examine the effects of video-assisted education about the intensive care process on intensive care experiences and anxiety levels of patients scheduled for open-heart surgery.

Research Hypotheses H01: Video-assisted education regarding the intensive care process provided to patients undergoing open heart surgery does not affect their experiences of intensive care.

H1: Video-assisted education regarding the intensive care process provided to patients undergoing open heart surgery does affect their experiences of intensive care.

H02: Video-assisted education regarding the intensive care process provided to patients undergoing open heart surgery does not affect patients' anxiety levels.

H2: Video-assisted education regarding the intensive care process provided to patients undergoing open heart surgery does affect patients' anxiety levels.

DETAILED DESCRIPTION:
The study will include an experimental and a control group. Patients in the experimental group will be administered the Patient Introduction Form, Trait Anxiety and State Anxiety Scales 48 hours before surgery. Then, video-assisted training will be given about the intensive care process, and the state anxiety scale will be applied again 24 hours before the surgery. Twenty-four hours after discharge from the intensive care unit to the clinic, the State Anxiety Scale and Intensive Care Experience Scales will be applied again. These scales will also be applied to patients in the control group who did not receive video-assisted education. Control group patients will not receive any intervention other than standard nursing care.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and over,
* Cognitively competent,
* Communicative and cooperative,
* Patients undergoing planned surgery (patients not admitted for emergency surgery),
* Patients without a psychiatric diagnosis,
* Patients with sensory impairments such as vision, hearing, or speech,
* Patients with stable hemodynamic status in the clinic,
* Patients who volunteered to participate in the study were included in the study.

Exclusion Criteria:

* Patients who did not volunteer to participate,
* Patients whose surgery was canceled,
* Patients who underwent emergency surgery,
* Patients who underwent combined bypass and valve surgery,
* Patients with previous intensive care experience,
* Patients who developed complications before, during, or after surgery were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Intensive care experience | 24 hours after arriving from intensive care care
  Intensive care experience will be evaluated with the Intensive Care Experience Scale. The scale has been developed to evaluate the experiences of patients in the intensive care unit.10 of the scale questions evaluate the frequency of the emotional condition in which the patient live, while the other 9 evaluate the compliance of the patient to intensive care. The substances prepared to evaluate the harmony of the patient in intensive care; Scored between 1 and 5.
Anxiety level | 48 hours before surgery, 24 hours before surgery, 24 hours after intensive care unit
  Anxiety level will be evaluated with the State-Trait Anxiety Inventory.The State-Trait Anxiety Inventory was first developed by Spielberger and colleagues in 1971, and its Turkish adaptation was completed by Öner and Le Compte in 1985. The scale consists of a total of 40 items and two separate subscales. The first 20 items assess individuals' state anxiety levels, while the remaining 20 items assess trait anxiety levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Atatürk University, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No